CLINICAL TRIAL: NCT03848923
Title: Impact of Thrombocytopenia and Platelet Transfusions on Neonatal Bleeding and Inflammation
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Martha Sola-Visner, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00029482; 2P01HL046925-21A1 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-02-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Thrombocytopenia
Keywords: Thrombocytopenia; Neonates; Platelets; NET Formation
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune; Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 study-specific blood samples (0.5-1.0 cc each) will be taken to the study laboratory for a CBC and plasma separation and storage for future measurements of dsDNA and MPO-DNA ELISA, markers of NET formation, TAT complexes (markers of intravascular coagulation), and for a panel of serum cytokines/vascular injury markers (IFNɣ, IL-6, IL-8, IL-10, IL-17, IL-18, TNFα/β, IP-10, MCP-1, ICAM, VCAM, and VEGF) by Luminex;
  In addition, left-over plasma samples from clinical tests will be collected daily from the clinical laboratory, aliquoted, and frozen for future cytokine measurements, as we did to generate the preliminary data for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study that was designed with the following two Specific Aims:

1. To determine whether the Immature Platelet Fraction percentage (IPF%) and the Immature Platelet Count (IPC) are better predictors of bleeding than the platelet count alone in neonates of different gestational and post-conceptional ages and with different etiologies of thrombocytopenia; and
2. To characterize the effects of neonatal thrombocytopenia and platelet transfusions (PLT Tx) on bleeding and on markers of systemic inflammation, thrombosis, and neutrophil extracellular traps (NET) formation in neonates with different underlying conditions.

DETAILED DESCRIPTION:
This is a prospective observational study designed to contrast the potential positive effects of neonatal platelet transfusion on clinical bleeding vs. their potentially negative effects on NET formation, intravascular thrombosis and elevation of pro-inflammatory cytokines.

Importantly, patients will be consented when they have a platelet count <100 x 109/L, but they will enter study only when the platelet count falls to <50 x 109/L.

After obtaining signed Informed Consent, enrolled infants will undergo the following:

1. Prospective collection of clinical and laboratory data, including:

1. Baseline demographic and clinical information from infants and mothers;
2. Clinical diagnoses at the time of enrollment (if NEC, then Bell's stage) and illness severity (SNAP scores) at the time of diagnosis;
3. All hemoglobins, hematocrits, PLT counts, IPF% and IPCs obtained during study. An IPF (the PLT equivalent of the reticulocyte count) is automatically run on every thrombocytopenic sample at all participating hospitals, and will provide information regarding mechanism of thrombocytopenia;
4. All blood culture results, and all markers of liver and renal function;
5. All PLT, RBC and plasma transfusions, including product characteristics, transfusion times, and volume; and
6. Neonatal outcomes including IVH (any grade), chronic lung disease (oxygen requirement at 36 wks post-conception), retinopathy of prematurity (any grade), and mortality.

Infants will be followed until resolution of the severe thrombocytopenia (PLT count >50x109/L without PLT Tx x 72 hours), death or discharge, whichever comes first.

2. Study-specific procedures. In addition to the data collected as above, enrolled infants will undergo the following study-specific measurements:

1. A bleeding score (Neo-BAT, see Appendix) will be obtained by the bedside nurse within 2 hours of every PLT count and IPF% checked. NeoBAT scores will include any bleeding since the last PLT count or over the prior 24 hours, whichever is shortest. This will serve to correlate bleeding scores with PLT counts, and to quantify changes following PLT Tx;
2. Two optional blood samples will be obtained within 2 hours prior to and 4±2 hours (see below) following the first clinically indicated PLT Tx after enrollment. These 2 study-specific blood samples (0.5-1.0 cc each) will be taken to the study laboratory for a CBC and plasma separation and storage for future measurements of dsDNA and MPO-DNA ELISA, markers of NET formation, TAT complexes (markers of intravascular coagulation), and for a panel of serum cytokines/vascular injury markers (IFNɣ, IL-6, IL-8, IL-10, IL-17, IL-18, TNFα/β, IP-10, MCP-1, ICAM, VCAM, and VEGF) by Luminex;
3. In addition, left-over plasma samples from clinical tests will be collected daily from the clinical laboratory, aliquoted, and frozen for future cytokine measurements, as we did to generate the preliminary data for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a post-menstrual age between 23 and 44 weeks;
2. Have a PLT count <100 x 109/L; and
3. Have a parent/guardian willing to provide written informed consent.

Exclusion Criteria:

1. Are not expected to survive for >5 days by the Attending Neonatologist;
2. Are thought to have a congenital thrombocytopenia or platelet dysfunction, based on family history or clinical presentation (e.g. congenital malformations, platelet morphology); or
3. Are on extracorporeal membrane oxygenation (ECMO).

Importantly, patients will be consented when they have a platelet count <100 x 109/L, but they will enter study only when the platelet count falls to <50 x 109/L.

Ages: 0 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will enroll neonates admitted to the NICUs at Boston Children's Hospital (BCH) and Beth Israel Deaconess Medical Center (BIDMC) and the Cardiac Intensive Care Unit (CICU) at BCH who fulfill the following criteria
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the bleeding score using the Neo-BAT (Neonatal Bleeding Assessment Tool), | Approximately 3 years
  The Neo-BAT categorizes bleeding as none (0), minor (1), moderate (2), severe (3), and major (4). A bleeding score will be obtained by the bedside nurse within 2 hours of every PLT count and IPF% checked. NeoBAT scores will include any bleeding since the last PLT count or over the prior 24 hours, whichever is shortest. This will serve to correlate bleeding scores with PLT counts, and to quantify changes following PLT Tx.

SECONDARY OUTCOMES:
Measurement of changes in cytokine levels and markers of intravascular coagulation and NET formation following PLT Tx | Approximately 3 years
  Cytokines will be measured within 2 hours before and 4 hours following a platelet transfusion using a Millipore multiplex immunoassay, analyzed with a BioPlex 200. All cytokine concentrations will be expressed in pg/mL. To measure NET formation at the same time points, we will use a newly described and validated ELISA to quantify citrullinated histone H3 (H3Cit) in plasma. This ELISA measures H3Cit in ng/mL. Increases in thrombin generation induced by platelet transfusions will be measured using a commercially available Thrombin-Antithrombin (TAT) Complex ELISA from Abcam, which measures TAT complexes in ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sola-Visner, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No